CLINICAL TRIAL: NCT01365091
Title: Bioequivalence Study of Fixed Dose Combinations of Saxagliptin/Metformin Extended Release (XR) Relative to Co-administration of the Individual Components in Healthy Subjects in the Fasted and Fed States
Brief Title: Bioequivalence Study of Fixed-dose Combinations and Coadministered Individual Tablets of Saxagliptin/Metformin-Brazil
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CV181-162
Record Dates: First submitted 2011-05-16; First posted 2011-06-03 (Estimated); Results first posted 2013-08-19 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1: Treatments A,B/B,A (Experimental): Period 1: Participants received a single oral dose of saxagliptin, 5 mg/metformin, 500 mg fixed-dose combination (FDC) in the fasted state (Treatment A), followed by a washout period of at least 7 days. Then, participants received single oral doses of saxagliptin, 5-mg, and metformin extended-release (XR), 500-mg, tablets together in the fasted state (Treatment B). Followed by a washout period of at least 4 days.
  Period 2: Participants received single oral doses of saxagliptin, 5-mg and metformin XR, 500-mg tablets together in the fasted state (Treatment B), followed by a washout period of at least 7 days. Then, participants received a single oral dose of saxagliptin, 5 mg/metformin, 500 mg FDC, in the fasted state (Treatment A).
  Interventions: Drug: Saxagliptin/metformin fixed-dose combination (FDC); Drug: Saxagliptin; Drug: Metformin extended-release (XR)
- Arm 2: Treatments C,D/D,C (Experimental): Period 1: Participants received a single oral dose of saxagliptin, 5 mg/metformin, 500 mg fixed-dose combination (FDC), in the fed state (Treatment C), followed by a washout period of at least 7 days. Then, participants received a single oral dose of saxagliptin, 5-mg, and metformin extended-release (XR), 500-mg tablets together in the fed state (Treatment D). Followed by a washout period of at least 4 days.
  Period 2: Participants received a single oral dose of saxagliptin, 5-mg and metforminXR, 500-mg tablets together in the fed state (Treatment D), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5 mg/metformin, 500 mg FDC, in the fed state (Treatment C).
  Interventions: Drug: Saxagliptin/metformin fixed-dose combination (FDC); Drug: Saxagliptin; Drug: Metformin extended-release (XR)
- Arm 3: Treatments E, F/F,E (Experimental): Period 1: Participants received a single oral dose of saxagliptin, 5 mg/metformin, 1000 mg fixed-dose combination (FDC), in the fasted state (Treatment E), followed by a washout period of at least 7 days. Participants received single oral doses of saxagliptin, 5-mg and metformin extended-release (XR), 1000-mg tablets together in the fasted state (Treatment F). Followed by a washout period of at least 4 days.
  Period 2: Participants received single oral doses of saxagliptin, 5- mg and metformin XR, 1000-mg tablets together in the fasted state (Treatment F), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5 mg/metformin, 1000 mg FDC, in the fasted state (Treatment E).
  Interventions: Drug: Saxagliptin; Drug: Saxagliptin/Metformin FDC; Drug: Metformin
- Arm 4: Treatments G,H/H,G (Experimental): Period 1: Participants received a single oral dose of saxagliptin , 5 mg/metformin, 1000 mg fixed-dose combination (FDC), in the fed state (Treatment G), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5-mg and metformin extended-release (XR), 1000-mg tablets together in the fed state (Treatment H). Followed by a washout period of at least 4 days.
  Period 2: Participants received a single oral dose of saxagliptin, 5-mg and metformin XR, 1000-mg tablets together in the fed state (Treatment H), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5 mg/metformin, 1000 mg FDC, in the fed state (Treatment G).
  Interventions: Drug: Saxagliptin; Drug: Saxagliptin/Metformin FDC; Drug: Metformin

INTERVENTIONS:
Drug: Saxagliptin/metformin fixed-dose combination (FDC) — Tablet, oral, 5 mg/500 mg FDC, once on Day 1 only, 1 day
  Other Names: Onglyza/Glucophage extended release (XR)
  Arms: Arm 1: Treatments A,B/B,A; Arm 2: Treatments C,D/D,C
Drug: Saxagliptin — Tablet, oral, 5 mg, once on Day 1 only, 1 day
  Other Names: Onglyza
Drug: Metformin extended-release (XR) — Tablet, oral, 500 mg, once on Day 1 only, 1 day
  Other Names: Glifage XR
  Arms: Arm 1: Treatments A,B/B,A; Arm 2: Treatments C,D/D,C
Drug: Saxagliptin/Metformin FDC — Tablet, Oral, 5 mg/1000 mg FDC, once on Day 1 only, 1 day
  Other Names: Onglyza/Glucophage XR
  Arms: Arm 3: Treatments E, F/F,E; Arm 4: Treatments G,H/H,G
Drug: Metformin — Tablet, oral, 1000 mg, once on Day 1 only, 1 day
  Other Names: Glifage XR
  Arms: Arm 3: Treatments E, F/F,E; Arm 4: Treatments G,H/H,G

SUMMARY:
To demonstrate the bioequivalence of saxagliptin and metformin in a saxagliptin, 5-mg/metformin extended-release (XR), 500-mg, fixed-dose combination (FDC) tablet with saxagliptin, 5-mg and metformin, 500-mg XR tablets administered together in both the fasted and fed states. In addition, to demonstrate the bioequivalence of saxagliptin and metformin in a saxagliptin, 5-mg/metformin XR, 1000-mg, FDC tablet with saxagliptin, 5-mg and metformin, 1000-mg XR tablets administered together in both the fasted and fed states.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy men and women
* women of childbearing potential who are using acceptable method of contraception
* Women who are not pregnant or nursing
* Body Mass Index (BMI) of 18 to 29.9 kg/m^2, inclusive. BMI=weight(kg)/height(m)^2.

Key Exclusion Criteria:

* Any significant acute or chronic medical illness.
* History of gastrointestinal (GI) disease
* Major surgery within 4 weeks of study drug administration
* Any GI surgery that could impact study drug absorption
* Donation of blood or plasma to a blood bank or in a clinical study (except a screening visit) within the 6 months of study drug administration.
* Blood transfusion within 3 months of study drug administration for women and within 2 months for men
* Inability to be venipunctured and/or tolerate venous access
* Current smoker or recent (within 1 month) history of regular tobacco use
* Recent (within 6 months of study drug administration) drug or alcohol abuse
* Participation in a bioequivalence study within the last 6 months of study drug administration
* Estimated creatinine clearance of <80 mL/min using Cockcroft-Gault formula
* History of allergy to drug class or related compounds
* History of allergy to metformin or other similar acting agents
* History of any significant drug allergy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2011-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Campinas, São Paulo, Brazil

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Treatments A/B, B/A: Period 1: Participants received a single oral dose of saxagliptin, 5 mg/metformin, 500 mg fixed-dose combination (FDC) in the fasted state (Treatment A), followed by a washout period of at least 7 days. Then, participants received single oral doses of saxagliptin, 5-mg, and metformin extended-release (XR), 500-mg, tablets together in the fasted state (Treatment B). Followed by a washout period of at least 4 days.
  Period 2: Participants received single oral doses of saxagliptin, 5-mg and metformin XR, 500-mg tablets together in the fasted state (Treatment B), followed by a washout period of at least 7 days. Then, participants received a single oral dose of saxagliptin, 5 mg/metformin, 500 mg FDC, in the fasted state (Treatment A).
- Arm 2: Treatments C/D, D/C: Period 1: Participants received a single oral dose of saxagliptin, 5 mg/metformin, 500 mg fixed-dose combination (FDC), in the fed state (Treatment C), followed by a washout period of at least 7 days. Then, participants received a single oral dose of saxagliptin, 5-mg, and metformin extended-release (XR), 500-mg tablets together in the fed state (Treatment D). Followed by a washout period of at least 4 days.
  Period 2: Participants received a single oral dose of saxagliptin, 5-mg and metforminXR, 500-mg tablets together in the fed state (Treatment D), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5 mg/metformin, 500 mg FDC, in the fed state (Treatment C).
- Arm 3:Treatments E/ F, F/E: Period 1: Participants received a single oral dose of saxagliptin, 5 mg/metformin, 1000 mg fixed-dose combination (FDC), in the fasted state (Treatment E), followed by a washout period of at least 7 days. Participants received single oral doses of saxagliptin, 5-mg and metformin extended-release (XR), 1000-mg tablets together in the fasted state (Treatment F). Followed by a washout period of at least 4 days.
  Period 2: Participants received single oral doses of saxagliptin, 5- mg and metformin XR, 1000-mg tablets together in the fasted state (Treatment F), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5 mg/metformin, 1000 mg FDC, in the fasted state (Treatment E).
- Arm 4: Treatments G/ H, H/G: Period 1: Participants received a single oral dose of saxagliptin , 5 mg/metformin, 1000 mg fixed-dose combination (FDC), in the fed state (Treatment G), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5-mg and metformin extended-release (XR), 1000-mg tablets together in the fed state (Treatment H). Followed by a washout period of at least 4 days.
  Period 2: Participants received a single oral dose of saxagliptin, 5-mg and metformin XR, 1000-mg tablets together in the fed state (Treatment H), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5 mg/metformin, 1000 mg FDC, in the fed state (Treatment G).
Period: Period 1
Arm/Group | Arm 1: Treatments A/B, B/A | Arm 2: Treatments C/D, D/C | Arm 3:Treatments E/ F, F/E | Arm 4: Treatments G/ H, H/G
Started | 28 | 28 | 28 | 28
Completed | 26 | 26 | 25 | 25
Not Completed | 2 | 2 | 3 | 3
Not completed — Adverse Event | 1 | 0 | 2 | 3
Not completed — Positive test result for drugs of abuse | 1 | 0 | 0 | 0
Not completed — No longer met study criteria | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Personal reasons | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Arm 1: Treatments A/B, B/A | Arm 2: Treatments C/D, D/C | Arm 3:Treatments E/ F, F/E | Arm 4: Treatments G/ H, H/G
Started | 26 | 26 | 25 | 25
Completed | 25 | 26 | 24 | 25
Not Completed | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Treatments A/B, B/A | Arm 2: Treatments C/D, D/C | Arm 3:Treatments E/ F, F/E | Arm 4: Treatments G/ H, H/G | Total
Number analyzed (Participants) | 28 | 28 | 28 | 28 | 112
Age, Customized [Number; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 55 years | 28 | 28 | 28 | 28 | 112
  >=55 years | 0 | 0 | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: Participants] — The clinical study report (CSR) stated only that participants of both genders were enrolled. The CSR did not report the number of each gender enrolled.
  Participants
    Both genders | 28 | 28 | 28 | 28 | 112

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentrations (Cmax) of Metformin, Saxagliptin, and 5-Hydroxy (5-OH) Saxagliptin as a Fixed-dose Combination (FDC) and as Individual Tablets
Time Frame: Days 1, 2, and 3 of Periods 1 and 2
Population: Participants who received study medication and were evaluable
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Sax, 5 mg/Met 500 mg XR FDC vs Individual Tablets, Fasted: Arm 1: Treatments A, B/B, A. Period 1: Participants received a single oral dose of saxagliptin (sax), 5-mg/metformin (met), 500-mg extended-release (XR) fixed-dose combination (FDC) in the fasted state (Treatment A), followed by a washout period of at least 7 days. Then, participants received single oral doses of saxagliptin, 5-mg, and metformin XR, 500-mg tablets together in the fasted state (Treatment B). Followed by a washout period of at least 4 days.
  Period 2: Participants received single oral doses of saxagliptin, 5-mg and metformin XR, 500-mg tablets together in the fasted state (Treatment B), followed by a washout period of at least 7 days. Then, participants received a single oral dose of saxagliptin, 5 mg/metformin, 500-mg FDC, in the fasted state (Treatment A).
- Sax, 5 mg/Met 500 mg vs FDC to Individual Tablets, Fed: Arm 2: Treatment C, D/D, C. Period 1: Participants received a single oral dose of saxagliptin (sax) 5-mg/metformin (met) 500-mg, extended-release (XR) fixed-dose combination (FDC), in the fed state (Treatment C), followed by a washout period of at least 7 days. Then, participants received a single oral dose of saxagliptin, 5-mg, and metformin XR, 500-mg tablets together in the fed state (Treatment D). Followed by a washout period of at least 4 days.
  Period 2: Participants received a single oral dose of saxagliptin, 5-mg and metformin XR, 500-mg tablets together in the fed state (Treatment D), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5-mg/metformin, 500-mg XR FDC, in the fed state (Treatment C).
- Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fasted: Arm 3: Treatment E, F/F, G. Period 1: Participants received a single oral dose of saxagliptin (sax), 5-mg/metformin (met), 1000-mg extended-release (XR) fixed-dose combination (FDC), in the fasted state (Treatment E), followed by a washout period of at least 7 days. Participants received single oral doses of saxagliptin, 5-mg, and metformin XR, 1000-mg tablets, together in the fasted state (Treatment F). Followed by a washout period of at least 4 days.
  Period 2: Participants received single oral doses of saxagliptin, 5-mg and metformin XR, 1000-mg tablets together in the fasted state (Treatment F), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5-mg/metformin, 1000-mg FDC, in the fasted state (Treatment E).
- Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fed: Arm 4: Treatments G,H/H,G. Period 1: Participants received a single oral dose of saxagliptin (sax), 5-mg/metformin (met), 1000-mg extended-release (XR) fixed-dose combination (FDC), in the fed state (Treatment G), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5-mg and metformin XR, 1000-mg tablets together in the fed state (Treatment H). Followed by a washout period of at least 4 days.
  Period 2: Participants received a single oral dose of saxagliptin, 5-mg and metformin XR, 1000-mg tablets together in the fed state (Treatment H), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5-mg/metformin, 1000-mg FDC, in the fed state (Treatment G).
Arm/Group | Sax, 5 mg/Met 500 mg XR FDC vs Individual Tablets, Fasted | Sax, 5 mg/Met 500 mg vs FDC to Individual Tablets, Fed | Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fasted | Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fed
Number analyzed (Participants) | 25 | 26 | 24 | 25
μg/mL
  Metformin Cmax (individual tablet) | 713 (176) [87.618 to 103.446] | 654 (118) [82.368 to 94.419] | 1177 (399) [90.376 to 105.404] | 1077 (139) [95.164 to 105.139]
  Metformin Cmax (FDC) | 678 (167) | 577 (95) | 1139 (325) | 1091 (214)
  Saxagliptin Cmax (individual tablet) | 29274 (10209) [96.552 to 119.924] | 28339 (7339) [92.263 to 104.451] | 30914 (7965) [96.956 to 109.407] | 31319 (6270) [89.055 to 98.470]
  Saxagliptin Cmax (FDC) | 31372 (11367) | 28140 (8311) | 33549 (7813) | 29545 (6006)
  5-OH Saxagliptin Cmax (individual tablets) | 54709 (16816) [96.504 to 112.883] | 52628 (12850) [91.470 to 98.714] | 56444 (14731) [96.589 to 108.52] | 55177 (13751) [95.572 to 103.144]
  5-OH Saxagliptin Cmax (FDC) | 56413 (15775) | 11316 (45404) | 59878 (15959) | 54521 (12319)
Statistical Analysis 1: Comparison: Sax, 5 mg/Met 500 mg XR FDC vs Individual Tablets, Fasted; Test type: Non-Inferiority or Equivalence — Metformin, Arm 1: The corresponding power and coefficient of variation between test and reference drugs are 98% and 17.24%, respectively; ANCOVA; Geometric mean ratio = 95.204, 90% CI 2-sided [87.618 to 103.446] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 2: Comparison: Sax, 5 mg/Met 500 mg XR FDC vs Individual Tablets, Fasted; Test type: Non-Inferiority or Equivalence — Saxagliptin, Arm 1: The corresponding power and coefficient of variation are 80% and 22.62%, respectively; ANCOVA; Geometric mean ratio = 107.606, 90% CI 2-sided [96.552 to 119.924] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 3: Comparison: Sax, 5 mg/Met 500 mg XR FDC vs Individual Tablets, Fasted; Test type: Non-Inferiority or Equivalence — 5-OH Saxagliptin, Arm 1: The corresponding power and the coefficient of variation are 99% and 16.26%, respectively; Geometric mean ratio = 104.373, 90% CI 2-sided [96.504 to 112.883] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B= FDC (test value)
Statistical Analysis 4: Comparison: Sax, 5 mg/Met 500 mg vs FDC to Individual Tablets, Fed; Test type: Non-Inferiority or Equivalence — Metformin, Arm 2: The corresponding power and the variation coefficient are 81% and 14.42%,respectively; ANCOVA; Geometric mean ratio = 88.188, 90% CI 2-sided [82.368 to 94.419] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 5: Comparison: Sax, 5 mg/Met 500 mg vs FDC to Individual Tablets, Fed; Test type: Non-Inferiority or Equivalence — Saxagliptin, Arm 2: The corresponding power and the variation coefficient are 99% and 13.09%, respectively; ANCOVA; Geometric mean ratio = 98.168, 90% CI 2-sided [92.263 to 104.451] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 6: Comparison: Sax, 5 mg/Met 500 mg vs FDC to Individual Tablets, Fed; Test type: Non-Inferiority or Equivalence — 5-OH saxagliptin, Arm 2: The corresponding power and the variation coefficient are 99% and 8.02%, respectively; ANCOVA; Geometric mean ratio = 95.023, 90% CI 2-sided [91.470 to 98.714] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 7: Comparison: Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fasted; Test type: Non-Inferiority or Equivalence — Metformin, Arm 3: The corresponding power and the variation coefficient are 99% and 15.55%, respectively; ANCOVA; Geometric mean ratio = 97.601, 90% CI 2-sided [15.55 to 99] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 8: Comparison: Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fasted; Test type: Non-Inferiority or Equivalence — Saxagliptin, Arm 3: The corresponding power and the variation coefficient are 84% and 15.65%, respectively; ANCOVA; Geometric mean ratio = 110.656, 90% CI 2-sided [102.416 to 119.559] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 9: Comparison: Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fasted; Test type: Non-Inferiority or Equivalence — OH-Saxagliptin, Arm 3: The corresponding power and the variation coefficient are 99% and 12.61%, respectively; ANCOVA; Geometric mean ratio = 106.264, 90% CI 2-sided [99.826 to 113.117] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 10: Comparison: Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fed; Test type: Non-Inferiority or Equivalence — Metformin, Arm 4: The corresponding power and the variation coefficient are 99% and 10.30%, respectively; ANCOVA; Geometric mean ratio = 100.028, 90% CI 2-sided [95.164 to 105.139] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 11: Comparison: Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fed; Test type: Non-Inferiority or Equivalence — Saxagliptin, Arm 4: The corresponding power and the variation coefficient are 99% and 10.38%, respectively; ANCOVA; Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value); Geometric mean ratio = 93.644, 95% CI 2-sided [89.055 to 98.470] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)

2. Primary Outcome: AUC From Time 0 to Time of the Last Quantifiable Concentration (AUC[0-T])of Metformin, Saxagliptin, and 5-Hydroxy (5-OH) Saxagliptin as a Fixed-dose Combination (FDC) and as Individual Tablets
Description: AUC=Area under the concentration-time curve
Time Frame: Days 1, 2, and 3 of Periods 1 and 2
Population: Participants who received study medication and were evaluable
Measure: Mean (Standard Deviation); unit: pg*h/mL
Groups:
- Sax, 5 mg/Met, 500 mg: Sax, 5 mg/Met, 500 mg FDC Fasting: Arm 1: Treatments A, B/B, A. Period 1: Participants received a single oral dose of saxagliptin (sax), 5-mg/metformin (met), 500-mg extended-release (XR) fixed-dose combination (FDC) in the fasted state (Treatment A), followed by a washout period of at least 7 days. Then, participants received single oral doses of saxagliptin, 5-mg, and metformin XR, 500-mg tablets together in the fasted state (Treatment B). Followed by a washout period of at least 4 days.
  Period 2: Participants received single oral doses of saxagliptin, 5-mg and metformin XR, 500-mg tablets together in the fasted state (Treatment B), followed by a washout period of at least 7 days. Then, participants received a single oral dose of saxagliptin, 5 mg/metformin, 500-mg FDC, in the fasted state (Treatment A).
- Sax, 5 mg/Met, 500 mg: Sax, 5 mg/Met 500 mg FDC Fed: Arm 2: Treatment C, D/D, C. Period 1: Participants received a single oral dose of saxagliptin (sax) 5-mg/metformin (met) 500-mg, extended-release (XR) fixed-dose combination (FDC), in the fed state (Treatment C), followed by a washout period of at least 7 days. Then, participants received a single oral dose of saxagliptin, 5-mg, and metformin XR, 500-mg tablets together in the fed state (Treatment D). Followed by a washout period of at least 4 days.
  Period 2: Participants received a single oral dose of saxagliptin, 5-mg and metformin XR, 500-mg tablets together in the fed state (Treatment D), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5-mg/metformin, 500-mg XR FDC, in the fed state (Treatment C).
- Sax, 5 mg/Met XR, 1000 mg: Sax, 5 mg/Met, 1000 mg FDC Fasting: Arm 3: Treatment E, F/F, G. Period 1: Participants received a single oral dose of saxagliptin (sax), 5-mg/metformin (met), 1000-mg extended-release (XR) fixed-dose combination (FDC), in the fasted state (Treatment E), followed by a washout period of at least 7 days. Participants received single oral doses of saxagliptin, 5-mg, and metformin XR, 1000-mg tablets, together in the fasted state (Treatment F). Followed by a washout period of at least 4 days.
  Period 2: Participants received single oral doses of saxagliptin, 5-mg and metformin XR, 1000-mg tablets together in the fasted state (Treatment F), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5-mg/metformin, 1000-mg FDC, in the fasted state (Treatment E).
- Sax, 5 mg/Met XR, 1000 mg: Sax, 5 mg/Met, 1000 mg FDC Fed: Arm 4: Treatments G,H/H,G. Period 1: Participants received a single oral dose of saxagliptin (sax), 5-mg/metformin (met), 1000-mg extended-release (XR) fixed-dose combination (FDC), in the fed state (Treatment G), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5-mg and metformin XR, 1000-mg tablets together in the fed state (Treatment H). Followed by a washout period of at least 4 days.
  Period 2: Participants received a single oral dose of saxagliptin, 5-mg and metformin XR, 1000-mg tablets together in the fed state (Treatment H), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5-mg/metformin, 1000-mg FDC, in the fed state (Treatment G).
Arm/Group | Sax, 5 mg/Met, 500 mg: Sax, 5 mg/Met, 500 mg FDC Fasting | Sax, 5 mg/Met, 500 mg: Sax, 5 mg/Met 500 mg FDC Fed | Sax, 5 mg/Met XR, 1000 mg: Sax, 5 mg/Met, 1000 mg FDC Fasting | Sax, 5 mg/Met XR, 1000 mg: Sax, 5 mg/Met, 1000 mg FDC Fed
Number analyzed (Participants) | 25 | 26 | 24 | 25
pg*h/mL
  Metformin AUC(0-T) (individual tablets) | 5816 (1859) [82.596 to 101.380] | 5071 (821) [85.560 to 98.035] | 8174 (2394) [96.956 to 109.407] | 9628 (3270) [85.502 to 101.053]
  Metformin AUC(0-T) (FDC) | 5386 (1896) | 4701 (1028) | 8500 (2713) | 8936 (2696)
  Saxagliptin AUC(0-T) (individual tablets) | 106070 (26733) | 110285 (22139) | 102913 (22067) | 124536 (24794) [98.494 to 104.147]
  Saxagliptin AUC(0-T) (FDC) | 103865 (31088) | 109345 (23947) | 99215 (20146) | 127232 (28709)
  5-OH Saxagliptin AUC(0-T) (individual tablets) | 320743 (68176) | 305354 (53254) | 324163 (59358) | 9628 (3270)
  5-OH Saxagliptin AUC(0-T) (FDC) | 331332 (67491) | 292515 (45404) | 323039 (56031) [96.512 to 103.648] | 8936 (2696) [97.367 to 102.932]
Statistical Analysis 1: Comparison: Sax, 5 mg/Met, 500 mg: Sax, 5 mg/Met, 500 mg FDC Fasting; Test type: Non-Inferiority or Equivalence — Metformin, Arm 1: The corresponding power and coefficient of variation are 98% and 17.24%, respectively; ANCOVA; Geometric mean ratio = 91.508, 90% CI 2-sided [82.596 to 101.380] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 2: Comparison: Sax, 5 mg/Met, 500 mg: Sax, 5 mg/Met, 500 mg FDC Fasting; Test type: Non-Inferiority or Equivalence — Saxagliptin, Arm 1: The corresponding power and the coefficient of variation are 99% and 07.66%, respectively; ANCOVA; Geometric mean ratio = 97.437, 90% CI 2-sided [93.889 to 101.119] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 3: Comparison: Sax, 5 mg/Met, 500 mg: Sax, 5 mg/Met, 500 mg FDC Fasting; Test type: Non-Inferiority or Equivalence — 5-OH Saxagliptin, Arm 1: The corresponding power and the coefficient of variation are 99% and 07.43%, respectively; ANCOVA; Geometric mean ratio = 96.770, 90% CI 2-sided [93.350 to 100.316] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 4: Comparison: Sax, 5 mg/Met, 500 mg: Sax, 5 mg/Met 500 mg FDC Fed; Test type: Non-Inferiority or Equivalence — Metformin, Arm 2: The corresponding power and the variation coefficient are 96% and 14.37%, respectively; ANCOVA; Geometric mean ratio = 91.585, 90% CI 2-sided [85.56 to 98.035] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 5: Comparison: Sax, 5 mg/Met, 500 mg: Sax, 5 mg/Met 500 mg FDC Fed; Test type: Non-Inferiority or Equivalence — Saxagliptin, Arm 2: The corresponding power and the variation coefficient are 96.028% and 101.095%, respectively; ANCOVA; Geometric mean ratio = 98.529, 90% CI 2-sided [96.028 to 101.095] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 6: Comparison: Sax, 5 mg/Met, 500 mg: Sax, 5 mg/Met 500 mg FDC Fed; Test type: Non-Inferiority or Equivalence — 5-OH Saxagliptin, Arm 2: The corresponding power and the variation coefficient are 99% and 6.55%, respectively; ANCOVA; Geometric mean ratio = 96.239, 90% CI 2-sided [93.286 to 99.286] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 7: Comparison: Sax, 5 mg/Met XR, 1000 mg: Sax, 5 mg/Met, 1000 mg FDC Fasting; Test type: Non-Inferiority or Equivalence — Metformin, Arm 3: The corresponding power and the variation coefficient are 99% and 12.19%, respectively; ANCOVA; Geometric mean ratio = 102.994, 90% CI 2-sided [96.956 to 109.407] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 8: Comparison: Sax, 5 mg/Met XR, 1000 mg: Sax, 5 mg/Met, 1000 mg FDC Fasting; Test type: Non-Inferiority or Equivalence — Saxagliptin, Arm 3: The corresponding power and the variation coefficient are 99% and 7.07%, respectively; ANCOVA; Geometric mean ratio = 97.135, 95% CI 2-sided [93.778 to 100.613] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 9: Comparison: Sax, 5 mg/Met XR, 1000 mg: Sax, 5 mg/Met, 1000 mg FDC Fasting; Test type: Non-Inferiority or Equivalence — 5-OH Saxagliptin, Arm 3: The corresponding power and the variation coefficient are 99% and 7.18%, respectively; ANCOVA; Geometric mean ratio = 100.01, 90% CI 2-sided [96.512 to 103.648] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 10: Comparison: Sax, 5 mg/Met XR, 1000 mg: Sax, 5 mg/Met, 1000 mg FDC Fed; Test type: Non-Inferiority or Equivalence — Metformin, Arm 1:The corresponding power and the variation coefficient are 93% and 17.35%, respectively; ANCOVA; Geometric mean ratio = 92.953, 90% CI 2-sided [85.502 to 101.053] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 11: Comparison: Sax, 5 mg/Met XR, 1000 mg: Sax, 5 mg/Met, 1000 mg FDC Fed; Test type: Non-Inferiority or Equivalence — Saxagliptin, Arm 4: The corresponding power and the variation coefficient are 99% and 5.75%, respectively; ANCOVA; Geometric mean ratio = 101.281, 95% CI 2-sided [98.494 to 104.147] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 12: Comparison: Sax, 5 mg/Met XR, 1000 mg: Sax, 5 mg/Met, 1000 mg FDC Fed; Test type: Non-Inferiority or Equivalence — 5-OH Saxagliptin, Arm 4: The corresponding power and the variation coefficient are 99% and 5.73%, respectively; ANCOVA; Geometric mean ratio = 100.111, 90% CI 2-sided [97.367 to 102.932] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)

3. Secondary Outcome: Number of Participants With Death as Outcome and Serious Adverse Events (SAEs)
Description: SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: Continuously, from screening through Day 1 to within 30 days of drug discontinuation on Day 1
Population: All enrolled participants who receive study medication
Measure: Number; unit: Participants
Groups:
- Arm 3: Treatments E,F/ F,E: Period 1: Participants received a single oral dose of saxagliptin, 5 mg/metformin, 1000 mg fixed-dose combination (FDC), in the fasted state (Treatment E), followed by a washout period of at least 7 days. Participants received single oral doses of saxagliptin, 5-mg and metformin extended-release (XR), 1000-mg tablets together in the fasted state (Treatment F). Followed by a washout period of at least 4 days.
  Period 2: Participants received single oral doses of saxagliptin, 5- mg and metformin XR, 1000-mg tablets together in the fasted state (Treatment F), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5 mg/metformin, 1000 mg FDC, in the fasted state (Treatment E).
- Arm 4: Treatments G,H/H,G: Period 1: Participants received a single oral dose of saxagliptin, 5 mg/metformin, 1000 mg fixed-dose combination (FDC), in the fed state (Treatment G), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5-mg and metformin extended-release (XR), 1000-mg tablets together in the fed state (Treatment H). Followed by a washout period of at least 4 days.
  Period 2: Participants received a single oral dose of saxagliptin, 5-mg and metformin XR, 1000-mg tablets together in the fed state (Treatment H), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5 mg/metformin, 1000 mg FDC, in the fed state (Treatment G).
Arm/Group | Arm 1: Treatments A,B/B,A | Arm 2: Treatments C,D/D,C | Arm 3: Treatments E,F/ F,E | Arm 4: Treatments G,H/H,G
Number analyzed (Participants) | 28 | 28 | 28 | 28
Participants
  Deaths | 0 | 0 | 0 | 0
  SAEs | 0 | 0 | 0 | 0

4. Primary Outcome: AUC From Time 0 Extrapolated to Infinite Time (AUC[0-inf]) for Metformin, Saxagliptin, and 5-Hydroxy (5-OH) Saxagliptin as a Fixed-dose Combination (FDC) and as Individual Tablets
Description: AUC=Area Under the Concentration-time Curve
Time Frame: Days 1, 2, and 3 of Periods 1 and 2
Population: Participants who received study medication and were evaluable
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Sax, 5 mg/Met 500 mg XR FDC to Individual Tablets, Fasted: Arm 1: Treatments A, B/B, A. Period 1: Participants received a single oral dose of saxagliptin (sax), 5-mg/metformin (met), 500-mg extended-release (XR) fixed-dose combination (FDC) in the fasted state (Treatment A), followed by a washout period of at least 7 days. Then, participants received single oral doses of saxagliptin, 5-mg, and metformin XR, 500-mg tablets together in the fasted state (Treatment B). Followed by a washout period of at least 4 days.
  Period 2: Participants received single oral doses of saxagliptin, 5-mg and metformin XR, 500-mg tablets together in the fasted state (Treatment B), followed by a washout period of at least 7 days. Then, participants received a single oral dose of saxagliptin, 5 mg/metformin, 500-mg FDC, in the fasted state (Treatment A).
- Sax, 5 mg/Met 500 mg XR FDC to Individual Tablets, Fed: Arm 2: Treatment C, D/D, C. Period 1: Participants received a single oral dose of saxagliptin (sax) 5-mg/metformin (met) 500-mg, extended-release (XR) fixed-dose combination (FDC), in the fed state (Treatment C), followed by a washout period of at least 7 days. Then, participants received a single oral dose of saxagliptin, 5-mg, and metformin XR, 500-mg tablets together in the fed state (Treatment D). Followed by a washout period of at least 4 days.
  Period 2: Participants received a single oral dose of saxagliptin, 5-mg and metformin XR, 500-mg tablets together in the fed state (Treatment D), followed by a washout period of at least 7 days. Participants received a single oral dose of saxagliptin, 5-mg/metformin, 500-mg XR FDC, in the fed state (Treatment C).
Arm/Group | Sax, 5 mg/Met 500 mg XR FDC to Individual Tablets, Fasted | Sax, 5 mg/Met 500 mg XR FDC to Individual Tablets, Fed | Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fasted | Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fed
Number analyzed (Participants) | 25 | 26 | 24 | 25
ng*h/mL
  Metformin AUC (0-inf) (individual tablets) | 5877 (1858) | 5127 (816) | 8338 (2414) | 9731 (3277)
  Metformin AUC (0-inf) (FDC) | 5443 (1905) [82.697 to 101.226] | 4754 (1037) [85.573 to 97.939] | 8618 (2726) [96.589 to 108.525] | 9054 (2684) [85.835 to 101.238]
  Saxagliptin AUC (0-inf) (individual tablets) | 107425 (26828) [93.955 to 101.132] | 111677 (22315) [96.044 to 101.090] | 104293 (22149) [93.832 to 100.662] | 125820 (24856) [98.574 to 104.196]
  Saxagliptin AUC (0-inf) (FDC) | 105248 (31314) | 110705 (24091) | 100620 (20264) | 128602 (28729)
  5-OH Saxagliptin AUC (0-inf) (individual tablets) | 337345 (67941) [93.393 to 100.247] | 310983 (53447) [93.319 to 99.290] | 330247 (59863) [96.560 to 103.594] | 332495 (62192) [97.324 to 102.864]
  5-OH Saxagliptin AUC (0-inf) (FDC) | 326501 (68475) | 298037 (45636) | 329085 (56298) | 332869 (59469)
Statistical Analysis 1: Comparison: Sax, 5 mg/Met 500 mg XR FDC to Individual Tablets, Fasted; Test type: Non-Inferiority or Equivalence — For AUC(0-inf) metformin, Arm 1, the corresponding power and coefficient of variation are 80% and 21.06%, respectively; ANCOVA; Geometric mean ratio = 91.494, 90% CI 2-sided [82.697 to 101.226] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 2: Comparison: Sax, 5 mg/Met 500 mg XR FDC to Individual Tablets, Fasted; Test type: Non-Inferiority or Equivalence — Saxagliptin, Arm 1: The corresponding power and the coefficient of variation are 99% and 07.60%, respectively; ANCOVA; Geometric mean ratio = 97.477, 90% CI 2-sided [93.955 to 101.132] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 3: Comparison: Sax, 5 mg/Met 500 mg XR FDC to Individual Tablets, Fasted; Test type: Non-Inferiority or Equivalence — 5-OH Saxagliptin, Arm 1. The corresponding power and the coefficient of variation are 99% and 07.31%, respectively; ANCOVA; Geometric mean ratio = 96.760, 90% CI 2-sided [93.393 to 100.247] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 4: Comparison: Sax, 5 mg/Met 500 mg XR FDC to Individual Tablets, Fed; Test type: Non-Inferiority or Equivalence — Metformin, Arm 2: The corresponding power and the variation coefficient are 96% and 14.25%, respectively; ANCOVA; Geometric mean ratio = 91.548, 90% CI 2-sided [85.573 to 97.939] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 5: Comparison: Sax, 5 mg/Met 500 mg XR FDC to Individual Tablets, Fed; Test type: Non-Inferiority or Equivalence — Saxagliptin, Arm 2: The corresponding power and the variation coefficient are 99% and 5.38%,respectively; ANCOVA; Geometric mean ratio = 98.535, 95% CI 2-sided [96.044 to 101.090] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 6: Comparison: Sax, 5 mg/Met 500 mg XR FDC to Individual Tablets, Fed; Test type: Non-Inferiority or Equivalence — 5-OH Saxagliptin, Arm 2: The corresponding power and the variation coefficient are 99% and 6.52%, respectively; ANCOVA; Geometric mean ratio = 96.258, 95% CI 2-sided [93.319 to 99.290] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 7: Comparison: Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fasted; Test type: Non-Inferiority or Equivalence — Metformin, Arm 3: The corresponding power and the variation coefficient are 99% and 11.75%, respectively; ANCOVA; Geometric mean ratio = 102.383, 95% CI 2-sided [96.589 to 108.525] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 8: Comparison: Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fasted; Test type: Non-Inferiority or Equivalence — Saxagliptin, Arm 5: The corresponding power and the variation coefficient are 99% and 7.07%, respectively; ANCOVA; Geometric mean ratio = 97.187, 90% CI 2-sided [93.832 to 100.662] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 9: Comparison: Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fasted; Test type: Non-Inferiority or Equivalence — 5-OH Sarexagliptin, Arm 3: The corresponding power and the variation coefficient are 99% and 7.08%, respectively; ANCOVA; Geometric mean ratio = 100.015, 95% CI 2-sided [96.560 to 103.594] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 10: Comparison: Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fasted vs Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fed; Test type: Non-Inferiority or Equivalence — Metformin, Arm 4: The corresponding power and the variation coefficient are 94% and 17.13%, respectively; ANCOVA; Geometric mean ratio = 93.219, 90% CI 2-sided [85.835 to 101.238]
Statistical Analysis 11: Comparison: Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fed; Test type: Non-Inferiority or Equivalence — Saxagliptin, Arm 4: The corresponding power and the variation coefficient are 99% and 5.72%, respectively; ANCOVA; Geometric mean ratio = 101.346, 90% CI 2-sided [98.574 to 104.196] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)
Statistical Analysis 12: Comparison: Sax, 5 mg/Met 1000 mg XR FDC to Individual Tablets, Fed; Test type: Non-Inferiority or Equivalence — 5-OH Saxagliptin, Arm 4: The corresponding power and the variation coefficient are 99% and 5.71%, respectively; ANCOVA; Geometric mean ratio = 100.056, 90% CI 2-sided [97.324 to 102.864] — Geometric mean ratio is calculated as B/A, where A=individual tablets (reference value) and B=FDC (test value)

ADVERSE EVENTS:
Time Frame: From screening through Day 1 to within 30 days of drug discontinuation on Day 1
Groups:
- Saxagliptin, 5 mg/Metformin XR, 1000 mg Fasting; Saxagliptin, 5 mg/Metformin XR, 1000 mg Fed; Saxagliptin, 5 mg/Metformin XR, 500 mg Fasting; Saxagliptin, 5 mg/Metformin XR, 500 mg Fed: XR=extended release
- Saxagliptin, 5 mg/Metformin, 1000 mg FDC Fasting; Saxagliptin, 5 mg/Metformin, 1000 mg FDC Fed; Saxagliptin, 5 mg/Metformin, 500 mg FDC Fasting; Saxagliptin, 5 mg/Metformin, 500 mg FDC Fed: FDC=fixed-dose combination
Arm/Group | Saxagliptin, 5 mg/Metformin XR, 1000 mg Fasting | Saxagliptin, 5 mg/Metformin XR, 1000 mg Fed | Saxagliptin, 5 mg/Metformin XR, 500 mg Fasting | Saxagliptin, 5 mg/Metformin XR, 500 mg Fed | Saxagliptin, 5 mg/Metformin, 1000 mg FDC Fasting | Saxagliptin, 5 mg/Metformin, 1000 mg FDC Fed | Saxagliptin, 5 mg/Metformin, 500 mg FDC Fasting | Saxagliptin, 5 mg/Metformin, 500 mg FDC Fed
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/28 | 0/28 | 0/28 | 0/28 | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 7/28 | 13/26 | 10/27 | 6/26 | 8/25 | 4/27 | 8/28 | 14/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Saxagliptin, 5 mg/Metformin XR, 1000 mg Fasting (N=28) | Saxagliptin, 5 mg/Metformin XR, 1000 mg Fed (N=26) | Saxagliptin, 5 mg/Metformin XR, 500 mg Fasting (N=27) | Saxagliptin, 5 mg/Metformin XR, 500 mg Fed (N=26) | Saxagliptin, 5 mg/Metformin, 1000 mg FDC Fasting (N=25) | Saxagliptin, 5 mg/Metformin, 1000 mg FDC Fed (N=27) | Saxagliptin, 5 mg/Metformin, 500 mg FDC Fasting (N=28) | Saxagliptin, 5 mg/Metformin, 500 mg FDC Fed (N=28)
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 1
White blood cell disorder (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Alanine aminotransferase abnormal (Investigations) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 10 | 1 | 4 | 2 | 7 | 4
Aptyalism (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Hypertension (Vascular disorders) | 1 | 3 | 0 | 1 | 0 | 1 | 2 | 1
Blood creatinine abnormal (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 6
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Red blood cell abnormality (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.